CLINICAL TRIAL: NCT06562543
Title: A Single Arm Phase 4 Trial to Evaluate the Safety and Efficacy of Oral Fruquintinib in the Treatment of Refractory Metastatic Colorectal Cancer in Patients From Minority Populations Underrepresented in Prior Fruquintinib Studies
Brief Title: A Trial to Evaluate the Safety and Activity of Fruquintinib in Minority Populations With Advanced, Previously Treated Colorectal Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-113-4002
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fruquintinib 5 mg (Experimental): Participants will receive fruquintinib capsule at a dose of 5 mg, orally (PO), once daily (QD), for the first 21 days of each 28-day treatment cycle until progressive disease (PD), unacceptable toxicity, or other discontinuation criteria are met.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Oral capsules
  Other Names: Fruzaqla™

SUMMARY:
High blood pressure (hypertension) is a known side effect of the treatment with fruquintinib. Current research does not provide a clear answer whether minority groups such as Black/African American and/or Hispanic/Latino with refractory metastatic colorectal cancer (mCRC) have a bigger risk of higher blood pressure after treatment with fruquintinib. The main aim of this study is to learn how often adults of a minority group experience hypertension after they have been treated with fruquintinib for refractory mCRC. Other aims are to learn how safe fruquintinib is and how well it is tolerated by participants.

Participants will receive fruquintinib in 4-week treatment cycles until their condition worsens, they do no longer tolerate the treatment or stop the treatment for other reasons. After the last treatment, participants will be checked upon every 3 months until study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written (or electronic) informed consent.
2. Male or female aged more than or equal to (≥)18 years.
3. Presence of histologically and/or cytologically documented metastatic colorectal adenocarcinoma. Rat sarcoma virus (RAS) status for each participant must be documented.
4. Have been previously treated with standard approved therapies:

   * Fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy,
   * An anti-vascular endothelial growth factor (VEGF) biological therapy (e.g., bevacizumab, aflibercept, ramucirumab [regorafenib is NOT an anti-VEGF biologic]), and
   * If RAS wild-type and medically appropriate, an anti-epidermal growth factor receptor (EGFR) therapy (e.g., cetuximab, panitumumab).
   * If known microsatellite instability-high (MSI-H) or deficient mismatch repair (dMMR) tumor and medically appropriate, a programmed cell death protein 1 (PD1) inhibitor.
5. Self-identify as Black and/or African American or Hispanic and/or Latino or as both.
6. Body weight ≥40 kilograms (kg).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at screening.
8. Have assessable disease according to RECIST version 1.1, assessed locally.
9. In participants of childbearing potential, agreement to use highly effective form(s) of contraception, which results in a low failure rate (less than [<]1 percent [%] per year) when used consistently and correctly, starting during the screening period, continuing throughout the entire trial period, and for 2 weeks after taking the last dose of the trial intervention. Such methods include oral (PO) hormonal contraception (combined estrogen/progestogen or progestogen-only) associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system (IUS), bilateral tubal ligation, vasectomized partner, or true sexual abstinence in line with the preferred and usual lifestyle of the participant. Those assigned male sex at birth must always use a condom.

Exclusion Criteria:

1. Absolute neutrophil count (ANC) <1.5 times 10^9 per liter (10^9/L), platelet count <100 times 10^9/L, or hemoglobin <9.0 grams per deciliter (g/dL). Blood transfusion within 1 week prior to enrollment for the purpose of increasing the likelihood of eligibility is not allowed.
2. Serum total bilirubin more than (>)1.5 times the upper limit of normal range (ULN). Participants with previously documented Gilbert syndrome and bilirubin <2 times ULN are eligible.
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times ULN in participants without hepatic metastases; ALT or AST >5 times ULN in participants with hepatic metastases.
4. Creatinine clearance <30 milliliters per minute (mL/min). Creatinine clearance can either be measured in a 24-hour urine collection or estimated by the Cockcroft-Gault equation. Where available and appropriate, other formulae may be used to estimate clearance after consultation with the trial medical monitor.
5. Urine dipstick or urinalysis with protein ≥2 positive or 24-hour urine protein ≥1.0 gram per 24 hours (g/24 hours). Participants with 1+ positive proteinuria must undergo a 24-hour urine collection to assess urine protein level.
6. Uncontrolled hypertension, defined as systolic BP ≥140 millimeter of mercury (mmHg) and/or diastolic blood pressure (BP) ≥90 mmHg despite optimal medical management. The participant must have BP below both limits. Repeated assessments are permitted.
7. International normalized ratio (INR) >1.5 times ULN or activated partial thromboplastin time (aPTT) >1.5 times ULN, unless the participant is currently receiving or intended to receive anticoagulants for prophylactic purposes.
8. History of or active gastric/duodenal ulcer or ulcerative colitis, active hemorrhage of an unresected gastrointestinal tumor, history of perforation or fistulas, or any other condition that could, in the investigator's judgment, result in gastrointestinal hemorrhage or perforation within the 6 months prior to screening.
9. History or presence of hemorrhage from any other site (e.g, hemoptysis or hematemesis) within 2 months prior to screening.
10. History of a thromboembolic event, including deep vein thrombosis, pulmonary embolism, or arterial embolism within 6 months prior to screening.
11. Stroke and/or transient ischemic attack within 12 months prior to screening.
12. Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction or coronary artery bypass surgery within 6 months prior to enrollment, severe or unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias requiring treatment, or left ventricular ejection fraction <50% by echocardiogram.
13. QT interval, corrected using the Fridericia method (QTcF) >480 milliseconds or any factors that increase the risk of QT interval, corrected based on the patient's heart rate (QTc) prolongation or risk of arrhythmic events such as hypokalemia, congenital long QT syndrome, or family history of long QT syndrome.
14. Systemic antineoplastic therapies (except for that described in exclusion criterion no. 15) or any investigational therapy within 2 weeks prior to the first dose of the trial intervention, including chemotherapy, radical radiotherapy, hormonotherapy, biotherapy, and immunotherapy.
15. Systemic small molecule targeted therapies (e.g., tyrosine kinase inhibitors [TKIs]) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of the trial intervention.
16. Palliative radiotherapy for bone metastasis/lesion within 2 weeks prior to the initiation of the trial intervention.
17. Brachytherapy (i.e., implantation of radioactive seeds) within 60 days prior to the first dose of the trial intervention.
18. Surgery or invasive procedure (i.e., a procedure that includes a biopsy; central venous catheter placement is allowed) within 14 days prior to the first dose of the trial intervention or unhealed surgical incision.
19. Any unresolved toxicities from previous antitumor treatments greater than NCI CTCAE, version 5.0, Grade 1 (except for alopecia or neurotoxicity Grade less than or equal to [≤]2).
20. Known human immunodeficiency virus infection.
21. Known history of active viral hepatitis. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load had to be undetectable on suppressive therapy, if indicated. Participants with hepatitis C virus (HCV) infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
22. Clinically uncontrolled active infection requiring intravenous (IV) antibiotics.
23. Tumor invasion of a large vascular structure (e.g., pulmonary artery or superior or inferior vena cava).
24. Those who are currently pregnant or lactating.
25. Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of SD for 14 days or longer; participants requiring steroids within 4 weeks prior to the start of the trial intervention are to be excluded.
26. Other malignancy, except for non-melanoma skin cancer, in situ cervical carcinoma, or bladder carcinoma (tumor in situ and T1) that had been adequately treated during the 5 years prior to screening. Participants with another primary malignancy that has been adequately treated may be included after consultation with the trial medical monitor.
27. Inability to take medication PO, dysphagia, or an active gastric ulcer resulting from previous surgery (e.g., gastric bypass) or a severe gastrointestinal disease, or any other condition that investigators believe might affect absorption of the investigational medicinal product (IMP).
28. Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition (e.g., current alcohol or drug abuse) that investigators suspect might prohibit use of the IMP, affect interpretation of trial results, or put the participant at undue risk of harm based on the investigator's assessment.
29. Known hypersensitivity to fruquintinib or any of its inactive ingredients, including the azo dyes Tartrazine- Federal Food, Drug, and Cosmetic Act (FD&C) Yellow 5 and Sunset yellow For Coloring Food (FCF)-FD&C Yellow 6.
30. Received prior fruquintinib.
31. Live vaccine ≤28 days before the first dose of the trial intervention. Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
32. Use of strong inducers of cytochrome P450 3A4 (CYP3A4) within 2 weeks before the first dose of the trial intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-10-04 (Estimated); Study Completion 2027-10-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Grade 3 and Grade 4 Hypertension | From the first dose of the study drug up to end of study (approximately 35 months)
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving the first dose of the study drug and within 30 days after the last dose of the study drug or the initiation of subsequent anti-cancer therapy, whichever occurs earlier. Severity (toxicity grade) for hypertension will be determined using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

SECONDARY OUTCOMES:
Number of Participants with TEAEs, Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and Deaths | From the first dose of the study drug up to end of study (approximately 35 months)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of the trial intervention. It does not necessarily have to have a causal relationship with trial intervention. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. An AESI is an AE of scientific and medical concern (including palmar-plantar erythrodysesthesia syndrome [hand-foot syndrome]) specific to the study drug or the same class of drugs (vascular endothelial growth factor [VEGF] inhibitors) for which ongoing monitoring and rapid communication by the investigator to Takeda may be appropriate. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect, or is considered medically significant event.
Overall Survival (OS) | Up to approximately 35 months
  OS will be defined as the interval from the first dose of fruquintinib until death.
Progression Free Survival (PFS) | Up to approximately 35 months
  PFS will be defined as the interval from the first dose of fruquintinib until the first radiographic documentation of objective progression assessed by investigator using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1, or death from any cause.
Confirmed Objective Response Rate (cORR) | Up to approximately 35 months
  Confirmed ORR is defined as the percentage of participants achieving a best overall response of confirmed complete response (CR) or partial response (PR), assessed by investigator per RECIST version 1.1. To be qualified for stable disease (SD), the duration of SD should last for at least 7 weeks.
Disease Control Rate (DCR) | Up to approximately 35 months
  DCR is defined as the percentage of participants achieving a best overall response of confirmed CR, PR, or SD, as assessed by investigator per RECIST version 1.1.
Duration of Response (DOR) | Up to approximately 35 months
  DOR is defined as the interval from the first occurrence of PR or CR, whichever comes first, until the date of radiographic PD or death. DOR will be determined for participants with the best overall response of confirmed CR or PR as assessed by investigator per RECIST version 1.1.
Plasma Concentration for Fruquintinib | Pre-dose (within 1 hour) on Day 21 of Cycles 1 and 2; 2 hours post-dose on Days 1 and 21 of Cycles 1 to 4 and 3 hours post-dose on Days 1 and 21 of Cycles 1 and 2 (cycle length=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- United States (44):
  - Central Alabama Research, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - PIH Health Whittier Hospital, Whittier, California
  - Christiana Care Health Services, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Baptist Health - Miami Cancer Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Indiana University, Indianapolis, Indiana
  - Our Lady of the Lake Physician Group - LSU Health Baton Rouge Oncology, Baton Rouge, Louisiana
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - MidAmerica Cancer Care, Kansas City, Missouri
  - SSM Health St. Louis DePaul Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Capital Health Medical Center - Hopewell, Pennington, New Jersey
  - Columbia University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - James J Peters Veterans Administration Medical Center - NAVREF, The Bronx, New York
  - Zangmeister Cancer Center, Columbus, Ohio
  - Hightower Clinical Research, Oklahoma City, Oklahoma
  - Jefferson Health, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center | Philadelphia, PA, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee -- Memphis, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Renovatio Clinical, El Paso, Texas
  - Oncology Consultants - Memorial City Location, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - BRCR Global, Katy, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Tranquil Research, Webster, Texas
  - UC Irvine Medical Center - Chao Family Comprehensive Cancer, Orange, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medstar Speciality Hospital, Northwest, Washington
- Fundacion de Investigacion de Diego (FDI Clinical Research), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/